CLINICAL TRIAL: NCT02556957
Title: CHWs, mHealth, and Combination HIV Prevention: An Implementation Science Cluster-Randomized Trial (mLAKE)
Brief Title: CHWs, mHealth, and Combination HIV Prevention
Acronym: mLAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00062089
Record Dates: First submitted 2015-09-20; First posted 2015-09-22 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2019-09

CONDITIONS: HIV
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HealthScouts Intervention (Experimental): HealthScouts (CHWs) regularly visit residents and counsel them using a motivational interviewing approach, supported by a smartphone application.
  Interventions: Behavioral: HealthScouts; Other: Standard of Care
- Standard of Care (Active Comparator): Referral by RCCS to HIV services. Free HIV clinic available in the community.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: HealthScouts
  Arms: HealthScouts Intervention
Other: Standard of Care

SUMMARY:
Kasensero, a fishing community on Lake Victoria in Uganda, is a representative HIV "hotspot" with extremely high HIV prevalence (44.3%) and incidence (~3.9/100py), yet low HIV service utilization. Hotspots such as Kasensero may seed and sustain HIV in general populations, compromising national and regional HIV control efforts. PEPFAR, UNAIDS, and WHO have recognized the urgent need to target hotspots with enhanced HIV treatment and prevention efforts. However, evidence on low-cost, comprehensive, and effective HIV control strategies for hotspots is limited and is thus a priority need for the field.

The investigators propose an implementation science, cluster-randomized, controlled trial in Kasensero to evaluate the impact on HIV service uptake and HIV incidence of CHWs promoting combination HIV prevention (CHP) services supported by mobile health technologies (mHealth). CHP is the implementation of multiple, evidence-based HIV prevention services (HIV testing and counseling, antiretroviral therapy, medical male circumcision, and behavior change) to maximize population-level impact on HIV incidence. For CHP to substantively decrease HIV incidence, most community members must be assessed for risk factors and current CHP utilization, then triaged, motivated, linked, and, if HIV-infected, retained in care. The proposed intervention will use low-cost CHWs leveraging mHealth decision support and counseling tools to promote CHP along this entire continuum of HIV service utilization. The hypotheses for this implementation science research are that residents in clusters receiving the implementation intervention will have improved CHP service uptake and decreased Population Prevalence of Viremia (PPDV) compared to controls receiving standard of care.

The intervention will be evaluated through a pragmatic, cluster-randomized trial nested within a large, ongoing population-based cohort study of HIV, the Rakai Community Cohort Study (RCCS). Intervention arm participants will be visited in their place of residence by CHWs trained to evaluate and triage participants into risk categories, provide tailored CHP health counseling, linkage, and adherence support, all supported by a mHealth decision support tool. The primary outcomes will be CHP service coverage and PPDV. Other outcomes will be HIV incidence, population viral load, implementation measures, retention, virologic suppression, and sexual behaviors.

Complimentary mixed methods (quantitative, qualitative, and cost) evaluations of the trial will be conducted to evaluate implementation processes, facilitators, and barriers to inform study results and future program uptake. Focus groups and in-depth interviews will be conducted during and after the follow-up period and synthesized with quantitative data. Intervention costs will be prospectively measured to provide information on program affordability.

Through this study, a novel, low-cost, and scalable implementation intervention to improve CHP uptake will be evaluated in an HIV "hotspot" critical to controlling the HIV epidemic. The study design ensures rigorous evidence of immediate relevance to many stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Kasensero

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3773 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Population Prevalence of Detectable Viremia | 4 Years
  Proportion of the entire population who have detectable HIV viremia
ART Coverage (self-report) | 4 Years
  Proportion of HIV+ persons who are on ART
HIV Care Coverage (self-report) | 4 years
  Proportion of HIV+ persons who are in HIV care
Medical Male Circumcision Coverage (self-report) | 4 years.
  Proportion of men who are circumcised

SECONDARY OUTCOMES:
HIV Incidence | 4 years.
Sexual Behaviors (self-report) | 4 years
  Proportion of the population which has multiple partners and/or inconsistent or no condom use
Population HIV Viral Load | 4 years
  The mean viral load of HIV+ persons
HIV Counseling and Testing Coverage (self-report) | 4 years
  Proportion of the entire population who have received HIV Counseling and Testing
HIV Prevalence | 4 years
  The prevalence of HIV in the entire population

CONTACTS AND LOCATIONS:
Overall Officials: Larry W Chang, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Rakai Health Sciences Program, Entebee, Uganda

REFERENCES:
- [Derived] Chang LW, Pollard R, Mbabali I, Anok A, Hutton H, Amico KR, Kong X, Mulamba J, Ssekasanvu J, Long A, Thomas AG, Thomas K, Bugos E, van Wickle K, Kennedy CE, Nalugoda F, Beres LK, Bollinger RC, Quinn TC, Serwadda D, Gray RH, Wawer MJ, Reynolds SJ, Nakigozi G. Mixed Methods, Implementation Science Evaluation of a Community Health Worker Strategy for HIV Service Engagement in Uganda. J Acquir Immune Defic Syndr. 2023 Sep 1;94(1):28-36. doi: 10.1097/QAI.0000000000003220. PMID 37195924
- [Derived] Chang LW, Mbabali I, Hutton H, Amico KR, Kong X, Mulamba J, Anok A, Ssekasanvu J, Long A, Thomas AG, Thomas K, Bugos E, Pollard R, van Wickle K, Kennedy CE, Nalugoda F, Serwadda D, Bollinger RC, Quinn TC, Reynolds SJ, Gray RH, Wawer MJ, Nakigozi G. Novel community health worker strategy for HIV service engagement in a hyperendemic community in Rakai, Uganda: A pragmatic, cluster-randomized trial. PLoS Med. 2021 Jan 6;18(1):e1003475. doi: 10.1371/journal.pmed.1003475. eCollection 2021 Jan. PMID 33406130
- [Derived] Chang LW, Mbabali I, Kong X, Hutton H, Amico KR, Kennedy CE, Nalugoda F, Serwadda D, Bollinger RC, Quinn TC, Reynolds SJ, Gray R, Wawer M, Nakigozi G. Impact of a community health worker HIV treatment and prevention intervention in an HIV hotspot fishing community in Rakai, Uganda (mLAKE): study protocol for a randomized controlled trial. Trials. 2017 Oct 23;18(1):494. doi: 10.1186/s13063-017-2243-6. PMID 29061194